CLINICAL TRIAL: NCT02188316
Title: The Histological Quality and Adequacy of Diminutive Colorectal Polyps Resected Using Jumbo Versus Hot Biopsy Forceps
Brief Title: Comparison of Jumbo and Hot Biopsy Forceps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camlıca Erdem Hospital (Other)
Responsible Party: Principal Investigator, Bulent Yasar, MD, Camlıca Erdem Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNEAH-KAEK 2014/22
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Colonoscopy; Polypectomy
Keywords: Cold forceps polypectomy; Diminutive colorectal polyp; Hot biopsy forceps electrocauterization; Jumbo forceps.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jumbo forceps polypectomy (Active Comparator): 89 patients were randomized to jumbo forceps arm and 120 diminutive colorectal polyps were removed by jumbo forceps polypectomy.
  Interventions: Device: Jumbo forceps
- Hot biopsy electrocauterization (Active Comparator): 90 patients were randomized to hot biopsy forceps arm and 117 diminutive colorectal polyps were removed by hot biopsy electrocauterization.
  Interventions: Device: Hot biopsy forceps

INTERVENTIONS:
Device: Jumbo forceps — comparison of different polypectomy devices
  Other Names: Jumbo forceps (Conmed, USA)
  Arms: Jumbo forceps polypectomy
Device: Hot biopsy forceps — comparison of different polypectomy devices
  Other Names: Hot biopsy forceps (Wilson-Cook Medical, USA)
  Arms: Hot biopsy electrocauterization

SUMMARY:
* Cold forceps polypectomy and hot biopsy forceps electrocauterization (HBF) are still widely used methods for endoscopic resection of diminutive colorectal polyps (DCPs)(polyps smaller than 5 mm). Jumbo forceps may be more effective in the removal of DCPs because of their larger size.
* This was a prospective study of consecutive patients undergoing colonoscopy and found to have at least one diminutive polyp. One experienced endoscopist removed DCPs using either jumbo or hot biopsy forceps.
* Aim was to evaluate the histological quality and adequacy of the DCPs resected using jumbo forceps in comparison with HBF.

DETAILED DESCRIPTION:
* Exclusion criteria were (i) having abnormal coagulation parameters and thrombocytopenia, taking aspirin or other medications which could affect bleeding time, (ii) history of inflammatory bowel disease, (iii) pregnancy.
* One experienced endoscopist carried out all the procedures using the same techniques.
* If a diminutive polyp was detected during colonoscopy, and it was estimated that the polyp was eligible for the study, the patient was randomly assigned by the physician to one of the two forceps groups (hot biopsy versus jumbo forceps) using a flipping coin method. Polypectomy was then performed with the intention to remove all polypoid tissue with one forceps bite. After the initial bite was obtained, the polypectomy site was observed with visual inspection. If residual polypoid tissue was observed after the first bite, additional biopsies were taken until visual eradication was attained.
* The size of the polyp was estimated during colonoscopy by visual comparison with the open biopsy forceps (Open-biopsy forceps technique). Polypectomies were performed using jumbo forceps (Conmed, USA) and hot biopsy forceps (Wilson-Cook Medical, USA). For HBF, the technique was based on the procedure first described in 1973, as follows: slight pulling force was applied to the polyp and then the electrocautery current was applied until the white coagulum was seen at the polyp base. The technique for jumbo forceps was as follows: after initial grasping, slight force was applied until the polyp was separated from the stalk. The electrocautery current waveform and intensity settings were the same for each patient. Each biopsy specimen was placed in a separate formalin solution.
* An experienced blinded pathologist evaluated the tissue samples for depth of specimen, amount of cautery damage (for hot biopsy forceps) or crush artifacts (for jumbo forceps), architecture, fragmentation, overall diagnostic quality, evaluation and positivity of surgical margins.
* All statistical analyses were performed using SPSS for Windows v. 15 (SPSS Inc., Chicago, IL, USA). Demographic, biochemical and histopathological features were classified as continuous or categorical variables. Kolmogorov-Smirnov analysis was used to test for Gaussian distribution. The data were expressed as arithmetic mean ± standard deviation (SD), since the evaluated variables were Gaussian-distributed. Comparisons between two groups were performed using the Student's t-test for continuous variables. Categorical variables were compared using the χ2 test (2X2, 3X2 and 4X2 tables) and Fisher's exact test. When the chi-square test was used, Yates' correction for continuity was used. All reported p-values were two-tailed, and those less than 0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients found to have at least one diminutive polyp (measuring ≤ 5 mm).

Exclusion Criteria:

* Having abnormal coagulation parameters and thrombocytopenia
* Taking aspirin or other medications which could affect bleeding time
* History of inflammatory bowel disease
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Complete eradication of diminutive polyps. | 3 months

SECONDARY OUTCOMES:
Adequate histopathological diagnosis | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Camlıca Erdem Hospital, Istanbul, Turkey (Türkiye)